CLINICAL TRIAL: NCT00306475
Title: Does The Addition Of Divalproex Sodium ER To An Atypical Antipsychotic Drug (APD) Improve Cognition And Psychopathology In Outpatients With Schizophrenia (SCH) Or Schizoaffective Disorder (SAD)?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other); Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 051231
Record Dates: First submitted 2006-03-22; First posted 2006-03-23 (Estimated); Results first posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2022-04

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: schizophrenia, cognition, mood stabilizer
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Divalproex Sodium Extended-Release Tablets
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Divalproex Sodium Extended-Release Tablets — divalproex sodium extended-release (ER) 1000 mg
  Arms: 1
Drug: placebo — placebo identical in appearance to active comparator
  Arms: 2

SUMMARY:
The major objective of this proposal is to test the hypothesis that the addition of divalproex sodium to an atypical antipsychotic drug other than clozapine will significantly improve: a) cognition; and b) psychopathology (positive, negative, and mood symptoms) in a double-blind, randomized trial of 6 weeks duration in patients with schizophrenia or schizoaffective disorder.

DETAILED DESCRIPTION:
Cognitive function is one of the most critical deficits in schizophrenia and schizoaffective disorder. It has been found that cognitive dysfunction may be even more important than positive or negative symptoms in predicting functional outcomes such as community adjustment, ability to work, social interactions, and caretaker burden. Preclinical data from our laboratory provided the rationale for a clinical trial to test whether divalproex sodium ER can improve cognitive impairment in patients.

The major objective of this proposal is to test the hypothesis that the addition of divalproex sodium to an atypical antipsychotic drug other than clozapine will significantly improve: a) cognition; and b) psychopathology (positive, negative, and mood symptoms) in a double-blind, randomized trial of 6 weeks duration in patients with schizophrenia or schizoaffective disorder.

ELIGIBILITY:
Inclusion criteria

* Male or female, age 18-65
* Diagnostic and Statistical Manual (DSM-IV) diagnosis of schizophrenia or schizoaffective disorder
* Treated with olanzapine, aripiprazole, ziprasidone, quetiapine or risperidone monotherapy for at least three months prior to enrollment
* Able to provide written consent

Exclusion criteria

* Primary DSM-IV diagnosis other than schizophrenia or schizoaffective disorder
* Treatment with any antipsychotic other than olanzapine, aripiprazole, ziprasidone, quetiapine or risperidone in the past three months
* Treatment with a mood stabilizer or an antidepressant continuously in the past three months. Patients who have had it for less than two weeks continuously will be permitted to enter.
* Pregnant or lactating females

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-03; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefania Bonaccorso, M.D., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Psychiatric Hospital at Vanderbilt, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Divalproex ER: Divalproex ER 500 mg/bid
- Placebo: Placebo 500 mg/bid
Period: Overall Study
Arm/Group | Divalproex ER | Placebo
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Divalproex ER: Divalproex 500 mgr ER
  Morning and Evening dose
  Active ingredient: Divalproex sodium
  500 mgr capsule by mouth. two times daily, one capsule in the morning and one capsule in the evening, for 6 weeks
- Placebo: Placebo
  Placebo: 2 capsules by mouth daily, one capsule in the morning and one capsule in the evening, for 6 weeks
- Total: Total of all reporting groups
Arm/Group | Divalproex ER | Placebo | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 60
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.93 (11.23) | 42 (10.0206) | 43.965 (10.7387571)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 29
  Male | 15 | 16 | 31
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Change in Cognition and Psychopathology Disorders as Measured on the MATRICS Consensus Cognitive Battery (MCCB)
Description: Giving Divalproex Sodium ER to Outpatients with Schizophrenia and Schizoaffective Disorder in addition to taking Atypical Antipsychotic Drug has shown to change their cognition and psychopathology.
  The MCCB measures cognitive function. The MCCB provides an overall composite score, expressed as a T-score, with a mean of 50 and a standard deviation of 10 The MCCB does not have minimum and maximum scores due to the use of T scores. A typical score will fall within a range of 40-60. Scores below 40 indicate impaired cognitive functioning, while scores above 60 suggest above-average cognitive abilities.
  The MCCB is often used in clinical research to assess cognitive deficits in individuals with psychiatric disorders, and the T-score scale is used to track cognitive changes over time.
Time Frame: six weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Participants Which Received IP: divalproex sodium extended-release (ER): divalproex sodium extended-release (ER) 1000 mg
- Participants Which Received Placebo: placebo identical in appearance to active comparator
Arm/Group | Participants Which Received IP | Participants Which Received Placebo
Number analyzed (Participants) | 30 | 30
units on a scale | 14.1 (2.8) | 14.3 (2.7)

ADVERSE EVENTS:
Groups:
- Divalproex Sodium: Active ingredient: Divalproex sodium ER: Divalproex sodium ER1000 mg. Assigned participants taking Divalproex sodium ER1000 mg in addition to their Atypical Antipsychotic Drug.
- Placebo: Placebo: Pill looks and tastes like the active ingredient but has no effect. Assigned participants taking Placebo in addition to their Atypical Antipsychotic Drug.
Arm/Group | Divalproex Sodium | Placebo
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Divalproex Sodium (N=30) | Placebo (N=30)
Any situation which makes the recurrence of severe Psychotic Symptoms, which is harmful to patients (General disorders) | 0 | 0
Severe Suicidal Ideation or suicidal attempt (Nervous system disorders) | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Divalproex Sodium (N=30) | Placebo (N=30)
Mild changes in patient's baseline state (General disorders) | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No